CLINICAL TRIAL: NCT05165810
Title: Evaluation of Multiple Interventions to Improve HIV Treatment Outcomes Among People Who Inject Drugs in India: a Randomized Factorial Trial With a Randomized Adaptive Component for Those Experiencing Early Treatment Failure
Brief Title: Evaluation of Multiple Interventions to Improve HIV Treatment Outcomes Among People Who Inject Drugs in India
Acronym: POINTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: YR Gaitonde Centre for AIDS Research and Education (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00232746; R01DA049301 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: People who inject drugs (PWID); Health services; Behavioral interventions; Antiretroviral Therapy; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This is a non-blinded, randomized, factorial trial with a secondary adaptive randomization, designed to assess the effectiveness of three interventions (relative to standard care) to increase viral suppression among HIV-positive PWID in India.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1: standard ART initiation + government-based HIV care + routine adherence support (Active Comparator): Participants randomized to Arm 1 will i) initiate ART on a standard timeline [usual care], ii) receive ongoing care in a government HIV clinic [usual care], and iii) receive routine adherence support should they experience treatment failure at 6 months [usual care].
  Interventions: Behavioral: Standard ART initiation [usual care]; Other: Government-based HIV care [usual care]; Behavioral: Routine adherence support [usual care]
- Arm 2: same-day ART + government-based HIV care + routine adherence support (Experimental): Participants randomized to Arm 2 will i) initiate ART on the day of enrollment [experimental], ii) receive ongoing care in a government HIV clinic [usual care], and iii) receive routine adherence support should they experience treatment failure at 6 months [usual care].
  Interventions: Behavioral: Same-day ART initiation [experimental]; Other: Government-based HIV care [usual care]; Behavioral: Routine adherence support [usual care]
- Arm 3: standard ART initiation + community-based HIV care + routine adherence support (Experimental): Participants randomized to Arm 3 will i) initiate ART on a standard timeline [usual care], ii) receive ongoing care in a PWID-focused community-based site [experimental], and iii) receive routine adherence support should they experience treatment failure at 6 months [usual care].
  Interventions: Behavioral: Standard ART initiation [usual care]; Other: Community-based HIV care [experimental]; Behavioral: Routine adherence support [usual care]
- Arm 4: standard ART initiation + government-based HIV care + enhanced adherence support (Experimental): Participants randomized to Arm 4 will i) initiate ART on a standard timeline [usual care], ii) receive ongoing care in a government HIV clinic [usual care], and iii) receive enhanced adherence support should they experience treatment failure at 6 months [experimental].
  Interventions: Behavioral: Standard ART initiation [usual care]; Other: Government-based HIV care [usual care]; Behavioral: Enhanced adherence support [experimental]
- Arm 5: same-day ART initiation + community-based-based HIV care + routine adherence support (Experimental): Participants randomized to Arm 5 will i) initiate ART on the day of enrollment [experimental], ii) receive ongoing care in a PWID-focused community-based site [experimental], and iii) receive routine adherence support should they experience treatment failure at 6 months [usual care].
  Interventions: Behavioral: Same-day ART initiation [experimental]; Other: Community-based HIV care [experimental]; Behavioral: Routine adherence support [usual care]
- Arm 6: same-day ART initiation + government-based-based HIV care + enhanced adherence support (Experimental): Participants randomized to Arm 6 will i) initiate ART on the day of enrollment [experimental], ii) receive ongoing care in a government HIV clinic [usual care], and iii) receive enhanced adherence support should they experience treatment failure at 6 months [experimental].
  Interventions: Behavioral: Same-day ART initiation [experimental]; Other: Government-based HIV care [usual care]; Behavioral: Enhanced adherence support [experimental]
- Arm 7: standard ART initiation + community-based-based HIV care + enhanced adherence support (Experimental): Participants randomized to Arm 7 will i) initiate ART on a standard timeline [usual care], ii) receive ongoing care in a PWID-focused community-based site [experimental], and iii) receive enhanced adherence support should they experience treatment failure at 6 months [experimental].
  Interventions: Behavioral: Standard ART initiation [usual care]; Other: Community-based HIV care [experimental]; Behavioral: Enhanced adherence support [experimental]
- Arm 8: same-day ART initiation + community-based-based HIV care + enhanced adherence support (Experimental): Participants randomized to Arm 8 will i) initiate ART on the day of enrollment [experimental], ii) receive ongoing care in a PWID-focused community-based site [experimental], and iii) receive enhanced adherence support should they experience treatment failure at 6 months [experimental].
  Interventions: Behavioral: Same-day ART initiation [experimental]; Other: Community-based HIV care [experimental]; Behavioral: Enhanced adherence support [experimental]

INTERVENTIONS:
Behavioral: Same-day ART initiation [experimental] — Participants assigned to same-day ART initiation will be offered standard, first-line ART on the day of trial enrollment. Participants, will be provided with focused counseling and instructions on where to follow-up for ongoing HIV care (either community-based HIV care or government-based HIV care, depending on randomization).
  Arms: Arm 2: same-day ART + government-based HIV care + routine adherence support; Arm 5: same-day ART initiation + community-based-based HIV care + routine adherence support; Arm 6: same-day ART initiation + government-based-based HIV care + enhanced adherence support; Arm 8: same-day ART initiation + community-based-based HIV care + enhanced adherence support
Behavioral: Standard ART initiation [usual care] — Participants randomized to standard ART initiation will not initiate ART on the day of trial enrollment, but only after linking to their assigned source of HIV care (either community-based HIV care or government-based HIV care, depending on randomization). In standard ART initiation, patients typically, complete an intake visit at the HIV clinic, with baseline laboratory testing, and return to the clinic approximately 2 weeks later to begin ART.
  Arms: Arm 1: standard ART initiation + government-based HIV care + routine adherence support; Arm 3: standard ART initiation + community-based HIV care + routine adherence support; Arm 4: standard ART initiation + government-based HIV care + enhanced adherence support; Arm 7: standard ART initiation + community-based-based HIV care + enhanced adherence support
Other: Community-based HIV care [experimental] — Participants randomized to community-based HIV care will be referred to PWID-focused integrated care centers (ICCs) for ongoing HIV clinical management - a prototype of decentralized HIV care in India. ICCs will provide free HIV care that will adhere closely to Indian HIV treatment guidelines and, when relevant, to local HIV treatment standards.
  Arms: Arm 3: standard ART initiation + community-based HIV care + routine adherence support; Arm 5: same-day ART initiation + community-based-based HIV care + routine adherence support; Arm 7: standard ART initiation + community-based-based HIV care + enhanced adherence support; Arm 8: same-day ART initiation + community-based-based HIV care + enhanced adherence support
Other: Government-based HIV care [usual care] — Participants randomized to government-based HIV care will be referred to government-based HIV clinics for ongoing HIV clinical management. Government-based clinics provide free HIV care that adheres closely to Indian HIV treatment guidelines
  Arms: Arm 1: standard ART initiation + government-based HIV care + routine adherence support; Arm 2: same-day ART + government-based HIV care + routine adherence support; Arm 4: standard ART initiation + government-based HIV care + enhanced adherence support; Arm 6: same-day ART initiation + government-based-based HIV care + enhanced adherence support
Behavioral: Enhanced adherence support [experimental] — Participants who i) experience virologic failure after 6 months in the study and ii) are randomized to enhanced adherence support will receive an intensive, tailored adherence intervention lasting a maximum of 6 months, with two components: 1) tracking and outreach, and 2) psychosocial support and navigation. These will aim to equip PWID with skills to independently manage their ART using motivational interviewing and strengths-based case management.
  Arms: Arm 4: standard ART initiation + government-based HIV care + enhanced adherence support; Arm 6: same-day ART initiation + government-based-based HIV care + enhanced adherence support; Arm 7: standard ART initiation + community-based-based HIV care + enhanced adherence support; Arm 8: same-day ART initiation + community-based-based HIV care + enhanced adherence support
Behavioral: Routine adherence support [usual care] — Participants who i) experience virologic failure after 6 months in the study and ii) are randomized to routine adherence support will receive a guideline-based, HIV clinic-based adherence counselling intervention lasting a maximum of 6 months
  Arms: Arm 1: standard ART initiation + government-based HIV care + routine adherence support; Arm 2: same-day ART + government-based HIV care + routine adherence support; Arm 3: standard ART initiation + community-based HIV care + routine adherence support; Arm 5: same-day ART initiation + community-based-based HIV care + routine adherence support

SUMMARY:
The goal of this study is to improve HIV care outcomes for people who inject drugs (PWID) in India. The study will implement a two-phase trial to evaluate whether HIV treatment outcomes (HIV viral suppression) in HIV infected PWID can be improved with three different interventions: i) by offering a faster treatment start time (same-day antiretroviral therapy [ART] initiation vs. standard), ii) by provided community-based HIV care in PWID-focused centers (vs. centralized government-based HIV care) and, iii) providing an enhanced adherence support to participants who experience treatment failure at six months (vs. routine adherence support). The investigators hypothesize that faster access to ART and HIV treatment in PWID-focused community sites will lead to higher levels of initiation and retention to ART compared with standard care; and use of enhanced navigation and psychosocial support to patients who experience treatment failure at six months will lead to improved viral suppression compared with routine adherence support.

DETAILED DESCRIPTION:
People who inject drugs (PWID) are at high risk for HIV infection and experience worse antiretroviral therapy (ART) outcomes than other key populations, particularly in low and middle income countries (LMIC). India has the largest number of opioid users in the world, and new injection drug epidemics have emerged in the North and Central regions of the country.

In phase 1, the investigators will evaluate two structural interventions to improve treatment outcomes among HIV-positive PWID in India. First, same-day ART (initiating ART on the day of HIV diagnosis/confirmation rather than waiting until standard evaluations are completed in an HIV clinic), was found to increase viral suppression rates in African studies with generalized HIV epidemics, but has not been evaluated in PWID. The second intervention is community-based HIV care. At present, all publicly-financed HIV treatment is provided at designated government ART centers. In prior work, the investigators found that PWID-centric integrated care centers (ICCs) were effective at engaging the population and increasing HIV testing uptake and were rated favorably by clients in anonymous surveys. ICCs linked HIV-positive PWID to government clinics, but were not equipped to provide primary HIV care. However, ICCs can be scaled-up to provide HIV treatment on-site and the investigators hypothesize this will improve initiation and retention to ART among PWID. The investigators will use a randomized factorial design to determine the individual and joint effects of same-day ART initiation and community-based HIV care. The primary outcome of the phase-1 trial is viral suppression at 6 months, with longer term follow-up to 18 months.

In phase 2, the investigators will evaluate a psychosocial/navigation intervention (enhanced adherence support) among participants who experience treatment failure during the first trial phase, defined as non-suppressed HIV RNA at the 6-month visit. These participants will be randomly assigned (in a second randomization) to enhanced adherence support or routine adherence support. The primary outcome of phase-2 will be viral suppression 6 months following the second randomization (12 months from enrollment in phase-1).

ELIGIBILITY:
PHASE 1 Inclusion Criteria:

* 18 years of age or older
* Reports injection drug use in prior 24 months
* Documented HIV positive
* Antiretroviral therapy naïve
* HIV RNA 1,000 c/mL or higher
* If previously linked to HIV care, able and willing to provide govt. ART book for documentation of care received.

PHASE 1 Exclusion Criteria:

* Pregnant (if female)
* Does not speak English, Hindi, or local language
* Plans to migrate in next 12 months
* Not competent to participate in the study or provide written informed consent.

PHASE 2 Inclusion Criteria:

• Participants who experience treatment failure at 6 months (HIV RNA>1000c/mL)

PHASE 2 Exclusion Criteria:

• Participants who do not experience treatment failure at 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with viral load suppression at 6 months after phase 1 randomization | Measured at 6 months after phase 1 randomization
  HIV RNA ≤1000 c/mL
Number of participants with viral load suppression at 12 months after phase 1 randomization | Measured at 6 months after the second randomization (12 months since phase 1 randomization)
  HIV RNA ≤1000 c/mL. Restricted to participants with treatment failure at 6 months who are allocated to either enhanced or routine adherence support in phase-2 randomization

SECONDARY OUTCOMES:
Number of participants with HIV viral suppression in each intervention at non-primary time points | Measured at 3, 12 and 18 months since phase 1 randomization
  HIV RNA ≤1000 c/mL
Mortality rate among participants | Measured at 3, 6, 12 and 18 months since phase 1 randomization
  To determine whether same-day ART, community HIV care, or enhanced adherence support affects mortality among HIV-positive PWID, relative to their control conditions.
Number of participants who are linked or re-linked (if in care previously) to HIV care | Measured up to 18 months after phase 1 randomization
  To determine whether same-day ART, community HIV care, or enhanced adherence support increases indices of the care continuum among HIV-positive PWID, relative to their control conditions.
Number of participants who initiate or re-initiate ART | Measured up to 18 months after phase 1 randomization
  To determine whether same-day ART, community HIV care, or enhanced adherence support increases indices of the care continuum among HIV-positive PWID, relative to their control conditions.
Number of participants who remain in HIV care | Measured up to 18 months after phase 1 randomization
  To determine whether same-day ART, community HIV care, or enhanced adherence support increases indices of the care continuum among HIV-positive PWID, relative to their control conditions.
Number of participants who adhere to their ART medication refills | Measured up to 18 months after phase 1 randomization
  To determine whether same-day ART, community HIV adherence support, or enhanced care increases indices of the care continuum among HIV-positive PWID, relative to their control conditions.
Number of participants who report increased quality of life since baseline | Measured at 3, 6, 12 and 18 months since phase 1 randomization
  Self-reported quality of life score based on amended version of validated instrument EQ-5D. To determine whether same-day ART, community HIV care, or enhanced adherence support increases quality of life (QOL) among HIV-positive PWID, relative to their control conditions.
Number of participants who engage with or are retained on medication for opioid use disorder (MOUD) | Measured at 3, 6, 12 and 18 months since phase 1 randomization
  To determine whether same-day ART, community HIV care, or enhanced adherence support increases use of and retention to medication for opioid use disorder (MOUD) among HIV-positive PWID, relative to their control conditions.
Number of participants who experience HIV-related stigma (anticipated, enacted, internalized) | Measured at 1, 3, 6, 12 and 18 months since phase 1 randomization
  Self-reported stigma scores based on 18-item likert scale

OTHER OUTCOMES:
Number of participants who develop antiretroviral drug resistance at follow-up compared with baseline | Measured at baseline, 3, 6, 12 and 18 months
  Measured using HIV-1 RNA-based genotyping assays.
Cost effectiveness analysis of providing each intervention relative to health outcomes | Measured from data captured across duration of trial up to five years
  Incremental cost-effectiveness ratios. Programmatic inputs will be measured separately and combined with prices (converted from local currency to US$) to generate total and per-client unit costs (e.g. average cost of patient enrolled). Unit prices for inputs will be obtained from financial records, itemized bills/receipts and sales catalogues. Personnel time will be costed by estimating time spent on intervention activities and apportioning salaries for staff in the market accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Lucas, PhD MD, Principal Investigator — Johns Hopkins University; Shruthi H Mehta, PhD MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- POINTER study -YRGCARE, New Delhi, India